CLINICAL TRIAL: NCT01373853
Title: A Single Centre Study to Compare the Efficacy and Safety of Femtosecond Laser-Assisted Versus Manual Cataract Surgery
Acronym: 1103
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1103
Record Dates: First submitted 2011-06-08; First posted 2011-06-15 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Cataract
Keywords: Lens Fragmentation; Cataract; Phacoemulsification; Femtosecond Laser
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femtec Groupe A (Experimental): In Group A the anterior capsulotomy and a pre-fragmentation of the ocular lens will be performed by means of femtosecond laser surgery
  Interventions: Procedure: Lens Fragmentation by means of a femtosecondlaser
- Manual Group B (Active Comparator): Group B acts as a control group where the capsulotomy and lens fragmentation are performed manually
  Interventions: Procedure: Manual Phacoemulsification

INTERVENTIONS:
Procedure: Lens Fragmentation by means of a femtosecondlaser — In Group A the anterior capsulotomy and a pre-fragmentation of the ocular lens will be performed by means of femtosecond laser surgery.
  Arms: Femtec Groupe A
Procedure: Manual Phacoemulsification — Group B acts as a control group where the capsulotomy and lens fragmentation are performed manually
  Arms: Manual Group B

SUMMARY:
This clinical study is a controlled, open, prospective, single-centre, multi-surgeon eye study to determine the safety and efficacy of intraocular cuts for femtosecond laser assisted lens frag-mentation to support phacoemulsification of the cataractous lens prior to IOL implantation. The cuts are applied by means of the FEMTEC femtosecond laser system with the CustomLens soft-ware module using a cylindrical and radial cut pattern with diameter and height dependent on anterior chamber depth, pupil diameter and ocular lens size.

The hypothesis of the study is that by means of femtosecond laser assisted lens fragmentation the required ultrasound energy used for phacoemulsification can be reduced in a safe and effective way.

ELIGIBILITY:
Inclusion Criteria:

* Clear corneal media
* Patients must be at least 18 years of age.

Exclusion Criteria:

* On a keratometric map of the cornea, the minimal and maximal K-values of the central 3mm zone must not differ by more than 5 dioptres. (exclusion criterium for Group A only)
* The maximum K- value may not exceed 60 D, the minimal value may not be smaller than 37 D. (exclusion criterium for Group A only)
* Corneal disease or pathology that precludes transmission of laser wavelength or distortion of laser light. (exclusion criterium for Group A only)
* Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally.
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye.
* Known sensitivity to planned concomitant medications.
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus
* Keratoconus
* Patients with woundhealing disorders such as connective tissue disease, autoimmune illnesses, immunodeficiency illnesses, ocular herpes zoster or simplex, endocrine diseases, lupus, rheumatoid arthritis
* Abnormal examination results from slit lamp, Fundus, IOL Master
* Abnormal examination results from Orbscan (exclusion criterium for Group A only)
* Patients with an autoimmune disease, collagenosis or clinically significant atopy.
* Patients who are pregnant or nursing.
* Patients who do not give informed consent.
* ACD < 2.4 mm or ACD > 4.5 mm as measured by ultrasonic examination (exclusion criterium for Group A only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Observation of the applied Effective Phaco Time (EPT) for Pahcoemulsifikation during surgery. The observed Effective Phaco Time in Group A should be significantly lower than in group B. Statistically significant difference at p<0.05. | at time of surgery

SECONDARY OUTCOMES:
Less or equal adverse events in Group A compared to group B (e.g. retinal detachment, IOL malposition). p<0.05 will be considered statistically significant. | 1-Day Follow-UP
Less or equal severe adverse events in Group A compared to group B. p<0.05 will be considered statistically significant. | 1-Day Follow-UP
Easy of phacoemulsification as subjectively perceived by the surgeon during surgery | time fo surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Maxivision Eye Hospital, Hyderabad, Andhra Pradesh, India